CLINICAL TRIAL: NCT06967116
Title: The Effect of Urinary Catheter Fixation on the Development of Meatal Pressure Injury in Male Patients Treated in Intensive Care Unit
Brief Title: Impact of Urinary Catheter Fixation on Meatal Pressure Injury in Male Patients in the Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merve Zorlu (Other)
Responsible Party: Sponsor-Investigator, Merve Zorlu, Nurse, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IU2024- 2948112
Record Dates: First submitted 2025-05-01; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-07

CONDITIONS: Urinary Catheter-Related Discomfort; Pressure Injury
Keywords: meatal pressure injury; fixation; intensive care; urinary catheter
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Using urinary catheter fixation tape) (Experimental): The area around the catheter entry point was cleaned twice a day during daytime (between 10.00-12.00) and evening (between 19.00-22.00) care hours of the unit and in case of additional need. On the first admission of the patient to the ICU, the urinary catheter was fixed to the leg with a fixation product and the catheter placement was changed to the other leg every 24 hours. The fixation product to be used fits every leg size thanks to its flexible structure and is securely fixed to the leg.
  Interventions: Procedure: Procedure Steps
- Control Group (standard care) (No Intervention): The area around the catheter entry point was cleaned during the daytime (10.00-12.00) and evening (19.00-22.00) maintenance hours of the unit and twice daily as needed.

INTERVENTIONS:
Procedure: Procedure Steps — The data of the study were collected with the 'Patient Identification Form' and 'Meatal Pressure Injury Daily Monitoring Form'.
  Arms: Experimental group (Using urinary catheter fixation tape)

SUMMARY:
Meatal pressure injury refers to the injury and ulceration of the head and shaft of the penis resulting from the constant pressure of an indwelling catheter. It can cause complications ranging from irritation and erythema of the skin and urethral epithelium to full-thickness tissue loss, penile deformity, and complete division of the penis, which may lead to sexual and urinary dysfunction. These complications can result in decreased quality of life and increased morbidity. Meatal pressure injury is a common problem in male patients in the ICU. However, studies on the prevention of meatal pressure injuries are very limited. This study is planned to evaluate the effectiveness of a urinary catheter fixation method on the development of meatal pressure injury in male patients treated in the intensive care unit.

DETAILED DESCRIPTION:
In this study, data were collected by the researcher from the hospital's electronic patient record system and by physical examination. Patients admitted to ICU were divided into two groups as experimental and control. The meatal pressure injury due to urinary catheter was determined by the investigator through physical examination. The first observation was made within the first 24 hours after the patient's admission to the clinic. During the physical examination, the patient's perineum was evaluated in terms of tissue integrity, moisture status, edema, lesions and redness and recorded by ensuring patient privacy. Physical examinations were performed by the researcher twice a day at the same time (08:00-09:00 in the morning and 20:00-21:00 in the evening). The data collection period was considered as 14 days. In case of meatal pressure injury, exitus, transfer of the patient to another unit, or removal of the urinary catheter, the data collection phase was terminated without waiting for the 14-day data collection follow-up period.

The study included 248 patients, 124 in the experimental group and 124 in the control group. Patients were randomly assigned to the experimental and control groups according to their sequence numbers. The study was designed as an open-label, randomized and controlled experimental study. A simple computer-assisted randomization method was used to ensure homogeneous group distribution. For this purpose, 248 sets were created using the functions available on the website "https://www.random.org/integer-sets".

The Meatal Pressure Injury Staging System developed by Shenhar (2020) categorizes injuries into four grades:

Grade 1 Meatal Pressure Injury: Erythematous, intact skin and mucosa. Grade 2 Meatal Pressure Injury: Partial loss of thick skin and mucosa. Grade 3 Meatal Pressure Injury: Less than 2 cm loss of full thickness skin and urethral mucosa.

Grade 4 Meatal Pressure Injury: Loss of 2 cm or more of full thickness skin and urethral mucosa.

In the study by Shenhar et al. these parameters were evaluated daily for two weeks. Permission to use the form was obtained from the responsible author.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Male patients in intensive care unit for at least 24 hours
* No existing meatal pressure injury
* Patients with urinary catheter on admission to the intensive care unit or urinary catheter inserted after intensive care unit admission

Exclusion Criteria:

* A skin disease that interferes with the assessment of pressure injury
* Any surgical intervention that prevents the evaluation of the meatal region
* Patients with condom urinary catheter

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since penis- related meatal pressure injury was evaluated in the study, male patients were included.
Enrollment: 248 (Actual)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Meatal Pressure Injury Staging System | Initial observation was made right after patient admission. Observations were repeated at 12-hour intervals for up to 14 days. Data collection was stopped earlier if a meatal pressure injury, death, transfer to another unit, or catheter removal occurred.
  Meatal Pressure Injury Staging System patients were monitored at 12 hour intervals. The patient's perineum and glans head were evaluated by observation. The staging system evaluates with 4 grades. These stages are as follows:
  * Grade 1: Meatus erosion is limited within the glans. Penile cleavage extends from the meatus to the proximal part of the cor-ona glans penis.
  * Grade 2: Erosion of the distal 1/3 of the penile shaft. Penile cleft extends from the meatus to the subcoronal part of the penis.
  * Grade 3: Erosion of the middle 1/3 of the penile shaft. Penile cleft extends from the meatus to the scrotum.
  * Grade 4: Erosion of the proximal 1/3 of the penile shaft/penoscrotal junction. The meatus is unaffected, but pressure necrosis is seen along the penile shaft.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Uslu, Assoc. Prof., Study Director — Istanbul University Nursinf Faculty
Locations (1):
- İstanbul University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The hypothesis results of the research will be shared. In this regard;
  * prevalence of meatal pressure injury
  * risk factors that increase meatal pressure injury

REFERENCES:
- [Background] Munien K, Ravichandran K, Flynn H, Shugg N, Flynn D, Chambers J, Desai D. Catheter-associated meatal pressure injuries (CAMPI) in patients with long-term urethral catheters-a cross-sectional study of 200 patients. Transl Androl Urol. 2024 Jan 31;13(1):42-52. doi: 10.21037/tau-23-445. Epub 2024 Jan 23. PMID 38404556
- [Background] Rassin M, Markovski I, Fishlov A, Naveh RU. An evaluation of preventing pressure ulcers in the urinary meatus. Dimens Crit Care Nurs. 2013 Mar-Apr;32(2):95-8. doi: 10.1097/DCC.0b013e31826bc65f. PMID 23388870
- [Background] Appah Y, Hunter KF, Moore KN. Securement of the Indwelling Urinary Catheter: A Prevalence Study. J Wound Ostomy Continence Nurs. 2016 Mar-Apr;43(2):173-7. doi: 10.1097/WON.0000000000000176. PMID 26418849
- [Background] Shenhar C, Mansvetov M, Baniel J, Golan S, Aharony S. Catheter-associated meatal pressure injury in hospitalized males. Neurourol Urodyn. 2020 Jun;39(5):1456-1463. doi: 10.1002/nau.24372. Epub 2020 Apr 27. PMID 32339318
- [Background] de Paula FM, Frota OP, Ruiz JS, Braulio IC, do Nascimento Goncalves FC, Ferreira-Junior MA, Sonobe HM, Ferreira DN, Pompeo CM, de Sousa AFL. Safety and efficacy of silicone tape for indwelling urinary catheter fixation in intensive care patients-A randomized clinical trial. Nurs Crit Care. 2024 Mar;29(2):347-356. doi: 10.1111/nicc.12937. Epub 2023 Jun 1. PMID 37264262
- [Background] Calpe-Damians N, Wennberg-Capellades L, Ventura-Rosado A, Gonzalez-Engroba R, Enriquez-Perez N, Vicario-Martos C, Roldos-Gales A, Guri-Lopez T, Rafart-Aguado S, Ramirez-Ramon A, Llaurado-Serra M. Effectiveness and safety of a simple catheter securement device aimed at preventing catheter-associated urinary tract infection in intensive care unit patients: A randomized controlled trial. Nurs Crit Care. 2024 Nov;29(6):1788-1798. doi: 10.1111/nicc.13111. Epub 2024 Jul 2. PMID 38955490